CLINICAL TRIAL: NCT00205075
Title: The Use of Validated Measures of Alcohol Intake to Measure the Impact of Moderate Alcohol Consumption on Hepatic Fibrogenesis in Individuals Infected With Hepatitis C
Brief Title: Impact of Moderate Alcohol Use on Hepatitis C Virus (HCV) Progression
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0161
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Hepatic Fibrogenesis; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Case
- Control

SUMMARY:
The purpose of this study is to determine the effect of moderate alcohol intake on liver disease caused by HCV in terms of speed of progression as compared to those not drinking alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with HCV who is not receiving or planning treatment but is receiving standard of care monitoring every 3 months and is either abstinent from alcohol or drinking only moderately

Exclusion Criteria:

* HIV co-infection
* Treated within the past 6 months
* History (hx) of other liver disease
* Alcohol use greater than 30 g/day or history of binge drinking in the last year
* Decompensated liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient with HCV not receiving or planning treatment but is receiving standard of care monitoring every 3 months, abstinent or drinking
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2004-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Said, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States